CLINICAL TRIAL: NCT00374244
Title: Efficacy of Pimozide Augmentation for Clozapine Partial Response
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02T-251
Record Dates: First submitted 2006-09-07; First posted 2006-09-11 (Estimated); Results first posted 2016-03-04 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-02

CONDITIONS: Schizophrenia
Keywords: schizophrenia; pimozide; clozapine
MeSH Terms: conditions — Schizophrenia | interventions — Pimozide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): placebo pimozide
  Interventions: Drug: placebo
- 2 (Active Comparator): active pimozide
  Interventions: Drug: Pimozide

INTERVENTIONS:
Drug: Pimozide — half of the subjects are randomized to the active drug group
  Arms: 2
Drug: placebo — half of the subjects are randomized to placebo group
  Arms: 1

SUMMARY:
This is a 12 week outpatient study for patients with schizophrenia who are on Clozapine, but continue to experience symptoms. The purpose of this project is to find out if small doses of pimozide (an antipsychotic medication, taken by mouth) will be helpful in reducing symptoms (such as hearing voices, having trouble in organizing your thoughts, lack of interest in life events and social activities), compared to placebo (an inactive substance, "sugar pill"), when added to clozapine in patients with schizophrenia.

The participant will be asked to come in once a week to meet with the research staff and study doctor. The participant will continue to see your regular clinician during this study for all normal appointments. The participant will remain on your current medications throughout the study. During the study you will be randomly selected to be put on a small dose of Pimozide or placebo.

DETAILED DESCRIPTION:
If you choose to participate, you will first have screening tests to find out if you are eligible. The study physician will do a number of tests including a physical examination, a routine medical history, lab tests for blood and urine, and EKG (to monitor your heart) and interviews about your physical and mental health.

At each visit you will complete an EKG (to monitor your heart), vital signs, and discuss how you are feeling with the research staff and doctor. Once a month, we will also conduct a slightly longer interview with you about your symptoms and draw one tube of blood to check your Clozapine level. At the beginning and end of the study, you will do some pencil and paper games called "Neurocognitive tests".

If you are interested in participating in this study, we will go over it in greater detail with you, including the possible benefits and risks associated with participating. We will make sure you understand the study before you begin. This study is completely voluntary, which means that you can choose to stop participating in the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder.
* A minimum Brief Psychiatric Rating Scale (BPRS) score of 35 and a BPRS psychotic symptom cluster score of at least 8.
* Currently taking clozapine with a blood level between 350-1000 ng/ml and on a stable dose of clozapine for the past 2 weeks.
* Able to give informed consent.

Exclusion Criteria:

* A history of significant medical/neurological disease such as thyroid, renal, hepatic abnormality, seizure disorder.
* History of Neuroleptic Malignant Syndrome.
* Current substance abuse determined by urine toxicology.
* Cardiac arrhythmia, sinus bradycardia (heart rate less than 60/min), sinus tachycardia (heart rate greater than 110/min), supraventricular tachycardia, ventricular tachycardia, Wolff-Parkinson-White Syndrome, first, second, third degree atrioventricular (AV) block, atrial fibrillation, atrial flutter and junctional complexes. in baseline electrocardiogram (EKG). Study doctors will examine the EKGs and consult with an internist/cardiologist as needed.
* on EKG: QTc > 450 ms.
* Current use of macrolide antibiotics (e.g., erythromycin, clarithromycin), azole antifungal agents (e.g., ketoconazole, itraconazole), protease inhibitors (e.g., ritonavir, indinavir), nefazodone, and other medications that are associated with prolonged QTc.
* Current use of antipsychotics other than clozapine.
* Current use of sertraline.
* IQ level below 70.
* At high risk for suicidal/homicidal behavior.
* Pregnancy, lack of birth control for females of childbearing age (female patients must report use of effective method for birth control such as birth control pills, condoms, barrier methods, abstinence or have written statement from their doctors that they are medically sterile).
* Non-English speaking.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2004-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Handan Gunduz-Bruce, MD, Principal Investigator — Yale University School of Medicine, Dept of Psychiatry
Locations (2):
- United States (2):
  - Connecticut Mental Health Center, New Haven, Connecticut
  - VA Connecticut Healthcare System, West Haven, Connecticut

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This clinical trial was conducted at the outpatient clinics of the West Haven VA, Connecticut Mental Health Center of Yale Department of Psychiatry, and the Zucker-Hillside Hospital of Long Island Jewish Health Care System, and approved by the respective Institutional Review Boards.
Pre-assignment Details: Prior to randomization, a stable dose of clozapine for the past 2 weeks with a blood level of at least 350 ng/ml was targeted. Subjects were stratified as to whether they were receiving psychoactive medications such as mood stabilizers, to ensure that about equal numbers of subjects were randomized based on this treatment profile.
Groups:
- Placebo Pimozide: Half of the subjects were randomized to placebo group.
- Active Pimozide: Half of the subjects are randomized to the active drug.
Period: Overall Study
Arm/Group | Placebo Pimozide | Active Pimozide
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Pimozide | Active Pimozide | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (2.8) | 44.3 (2.0) | 43.0 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Brief Psychiatric Rating Scale (BPRS) Total Score
Description: The Brief Psychiatric Rating Scale (BPRS) is an 18-item instrument. The items are anchored on a 7-point scale (higher rating: greater severity). Total scores range from 18 to 126 (higher score: greater severity). The instrument covers areas including: somatic concerns, anxiety, emotional withdrawal, conceptual disorganization, guilt feelings, tension, mannerisms and posturing, grandiosity, depressive mood, hostility, suspiciousness, hallucinatory behavior, motor retardation, uncooperativeness, unusual thought content, blunted affect, excitement and disorientation.
Time Frame: Baseline
Population: Subjects were analyzed intent to treat.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Pimozide | Active Pimozide
Number analyzed (Participants) | 14 | 14
units on a scale | 44.1 (2.0) | 44.3 (2.0)

2. Primary Outcome: Brief Psychiatric Rating Scale (BPRS) Total Score
Description: as for outcome 1
Time Frame: Endpoint (12 weeks)
Population: Subjects were analyzed intent to treat.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Pimozide | Active Pimozide
Number analyzed (Participants) | 14 | 14
units on a scale | 37.9 (2.1) | 39.6 (2.1)

3. Secondary Outcome: CGI Severity of Illness Scale (CGI-S)
Description: CGI Severity of Illness Scale (CGI-S) assesses severity of illness on 1-7 scale. Clinicians' experience is used to gauge the severity of illness from 'normal' (value=1) to 'among the most extremely ill patients' (value=7). The higher rating correlates with more severely ill.
Time Frame: baseline
Population: Analyzes intent to treat.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Pimozide | Active Pimozide
Number analyzed (Participants) | 14 | 14
units on a scale | 4.1 (0.5) | 4.0 (0.9)

4. Secondary Outcome: CGI Severity of Illness Scale (CGI-S)
Description: as for outcome 3
Time Frame: Endpoint (12 weeks)
Population: Analyzed intent to treat.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Pimozide | Active Pimozide
Number analyzed (Participants) | 14 | 14
units on a scale | 3.9 (0.8) | 3.9 (0.5)

5. Secondary Outcome: CGI Improvement Scale (CGI-I)
Description: CGI Improvement Scale (CGI-I) higher rating correlates with worsening of condition (vs. improvement with lower rating). The CGI-I is scored from 1 to 7 where 1 = 'very much improved' and 7 = 'very much worse'. Clinicians are asked to rate total improvement in the following manner: "...in your judgement, it is due entirely to drug treatment. Compared to his condition at admission to the project, how much has he changed?"
Time Frame: Endpoint (12 weeks)
Population: Analyzed intent to treat.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Pimozide | Active Pimozide
Number analyzed (Participants) | 14 | 14
units on a scale | 2.8 (1.0) | 3.4 (0.5)

6. Primary Outcome: Scale for the Assessment of Negative Symptoms (SANS)
Description: The Scale for the Assessment of Negative Symptoms (SANS) is a rating scale to measure negative symptoms in schizophrenia. The scale has 25 items (20 individual and 5 global) rated on scale of 0-5 (higher rating: greater severity). SANS is split into 5 domains, and within each domain separate symptoms are rated from 0 (absent) to 5 (severe). Domains include: Affective Flattening or Blunting, Alogia, Avolition - Apathy, Anhedonia - Asociality, Attention. The total range of the SANS is from 0 to 120.
Time Frame: baseline
Population: Analyzed intent to treat.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Pimozide | Active Pimozide
Number analyzed (Participants) | 14 | 14
units on a scale | 44.3 (5.9) | 38.5 (5.8)

7. Primary Outcome: Scale for the Assessment of Negative Symptoms (SANS)
Description: as for outcome 6
Time Frame: Endpoint (12 weeks)
Population: Analyzed intent to treat.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Pimozide | Active Pimozide
Number analyzed (Participants) | 14 | 14
units on a scale | 36.3 (5.9) | 37.3 (5.9)

8. Secondary Outcome: Verbal Fluency
Description: Verbal fluency was measured using the Controlled Word Association Test (COWAT). There is no range for this measure, as it is not a scale. The subjects can generate as many new words as they can, so there is no maximum. The greater the number of words one generates indicates better performance.
Time Frame: Baseline
Population: Intent to Treat Analysis
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Placebo Pimozide | Active Pimozide
Number analyzed (Participants) | 14 | 14
words | 12.2 (1.4) | 10.5 (1.5)

9. Secondary Outcome: Verbal Fluency
Description: as for outcome 8
Time Frame: Endpoint (12 weeks)
Population: Intent to Treat Analysis
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Placebo Pimozide | Active Pimozide
Number analyzed (Participants) | 14 | 14
words | 12.3 (1.5) | 11.1 (1.5)

10. Secondary Outcome: QTc
Description: The QT interval is a measure of the time between the start of the Q wave and the end of the T wave in the heart. ECG machines calculate a corrected QT (QTc). QTc is the corrected QT interval in the EKG. Normal range is from 430-470ms.
Time Frame: Baseline
Population: Intention to Treat
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo Pimozide | Active Pimozide
Number analyzed (Participants) | 14 | 14
ms | 408.8 (5.0) | 412.3 (5.1)

11. Secondary Outcome: QTc
Description: as for outcome 10
Time Frame: Endpoint (12 weeks)
Population: Intention to Treat
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo Pimozide | Active Pimozide
Number analyzed (Participants) | 14 | 14
ms | 412.9 (5.0) | 420.3 (5.2)

12. Secondary Outcome: Processing Speed
Description: Processing speed was assessed using using Digit Symbol Coding from the Wechsler Adult Intelligence Scale, Revised (WAIS-R). The tool is used for the assessment of processing speed. The range of scores is 0 to 100- with the higher number indicating greater performance.
Time Frame: Baseline
Population: Intent to Treat Analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Pimozide | Active Pimozide
Number analyzed (Participants) | 14 | 14
units on a scale | 48.8 (4.6) | 43.3 (4.9)

13. Secondary Outcome: Processing Speed
Description: as for outcome 12
Time Frame: Endpoint (12 weeks)
Population: Intent to Treat Analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Pimozide | Active Pimozide
Number analyzed (Participants) | 14 | 14
units on a scale | 46.5 (4.7) | 42.8 (5.0)

14. Secondary Outcome: Verbal Learning and Memory: List A
Description: Verbal learning and memory were assessed by the Rey Auditory Verbal Learning Test (RAVLT) List A: Total Trials (1-5). This assessment consists of a list of words that the subject repeats back, it does not have an interpret-able range of scores like a traditional scale. Scores are based on number of words repeated back.
Time Frame: Baseline
Population: Intent to Treat Analysis
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Placebo Pimozide | Active Pimozide
Number analyzed (Participants) | 14 | 14
words | 40.0 (3.3) | 26.5 (2.8)

15. Secondary Outcome: Verbal Learning and Memory: List A
Description: as for outcome 14
Time Frame: Endpoint (12 weeks)
Population: Intent to Treat Analysis
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Placebo Pimozide | Active Pimozide
Number analyzed (Participants) | 14 | 14
words | 38.0 (4.8) | 32.3 (4.2)

16. Secondary Outcome: Verbal Learning and Memory: List B
Description: Verbal learning and memory were assessed by the Rey Auditory Verbal Learning Test (RAVLT) List B: Single Trial. This assessment consists of a list of words that the subject repeats back, it does not have an interpret-able range of scores like a traditional scale. Scores are based on number of words repeated back.
Time Frame: Baseline
Population: Intent to Treat Analysis
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Placebo Pimozide | Active Pimozide
Number analyzed (Participants) | 14 | 14
words | 3.8 (0.4) | 3.5 (0.4)

17. Secondary Outcome: Verbal Learning and Memory: List B
Description: as for outcome 16
Time Frame: Endpoint (12 weeks)
Population: Intent to Treat Analysis
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Placebo Pimozide | Active Pimozide
Number analyzed (Participants) | 14 | 14
words | 3.4 (0.6) | 3.9 (0.6)

18. Secondary Outcome: Trail Making Test: Trail A
Description: Working memory by Digit Span and Letter Number Sequencing, and attention/executive functions were measured by the Trail Making Test (Parts A and B). This is an assessment of attention/executive function, it does not have an interpret-able range of scores like a traditional scale. Subjects makes trails on paper against time.
Time Frame: Baseline
Population: Intent to Treat Analysis
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo Pimozide | Active Pimozide
Number analyzed (Participants) | 14 | 14
seconds | 3.7 (0.1) | 3.8 (0.1)

19. Secondary Outcome: Trail Making Test: Trail A
Description: The Trail Making Test is a neuropsychological test of visual attention and task switching. It consists of two parts in which the subject is instructed to connect a set of 25 dots as fast as possible while still maintaining accuracy. ( Arnett, James A.; Seth S. Labovitz (1995). "Effect of physical layout in performance of the Trail Making Test". Psychological Assessment 7 (2): 220-221. doi:10.1037/1040-3590.7.2.220. Retrieved 2012-02-22.)
  Part A is used primarily to examine cognitive processing speed. Part B, in which the subject alternates between numbers and letters, is used to examine executive functioning. (Tombaugh, T.N.T.N (2004). "Trail Making test A and B: Normative Data Stratified by Age and Education". Archives of Clinical Neuropsychology : The Official Journal of the National Academy of Neuropsychologists 19 (2): 203-214. doi:10.1016/s0887-6177(03)00039-8. Retrieved 2012-01-10.)
Time Frame: Endpoint (12 weeks)
Population: Intent to Treat Analysis
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo Pimozide | Active Pimozide
Number analyzed (Participants) | 14 | 14
seconds | 3.6 (0.1) | 3.8 (0.1)

20. Secondary Outcome: Trail Making Test: Trail B
Description: as for outcome 19
Time Frame: Baseline
Population: Intent to Treat Analysis
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo Pimozide | Active Pimozide
Number analyzed (Participants) | 14 | 14
seconds | 4.6 (0.2) | 4.9 (0.2)

21. Secondary Outcome: Trail Making Test: Trail B
Description: as for outcome 19
Time Frame: Endpoint (12 weeks)
Population: Intent to Treat Analysis
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo Pimozide | Active Pimozide
Number analyzed (Participants) | 14 | 14
seconds | 4.6 (0.2) | 4.9 (0.2)

ADVERSE EVENTS:
Arm/Group | Placebo Pimozide | Active Pimozide
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 1/14 | 1/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Pimozide (N=14) | Active Pimozide (N=14)
QTc Prolongation (Cardiac disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No